CLINICAL TRIAL: NCT01876667
Title: An Evaluation of Clinical Pharmacist-led Intervention on Clinical Outcomes in Patients With Ischemic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPCRS stroke study; 10010533 - KPCO IRB (Other: KPCO)
Record Dates: First submitted 2012-08-28; First posted 2013-06-12 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Methods; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (CPCRS) Group (Active Comparator): CPCRS will ensure patients have regular laboratory monitoring and blood pressure measures, appropriate lipid-lowering and antihypertensive medications, and receive follow-up in a timely manner.
  Interventions: Other: Intervention (CPCRS) Group
- Usual Care (Placebo Comparator): Usual Care: Patients randomized to Usual Care will continue to receive interventions/procedures they normally receive according to standard/usual care practices
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Intervention (CPCRS) Group — CPCRS staff will order evidence-based lipid-lowering and/or antihypertensive medications, adjust doses, and order follow-up laboratory parameters, as necessary under pre-approved regional treatment protocols. Patients will be monitored for medication adherence and adverse effects. Patients receive dietary, exercise, and smoking cessation counseling verbally and through mailing of pre-printed Kaiser Permanente approved, patient education pamphlets, as necessary per the discretion of the clinical pharmacy specialist. Patients requiring more dietary counseling will be referred to dieticians, education classes, or other appropriate resources offered at KPCO. Primary care providers will be informed of all medication initiations or dosage adjustments.
  Arms: Intervention (CPCRS) Group
Other: Placebo — Usual Care
  Arms: Usual Care

SUMMARY:
Clinical pharmacy specialists are in an ideal position to assist medical teams in the management of patients with ischemic stroke. Given their extensive and specialized knowledge regarding medication efficacy, safety, and cost-effective use as well as their ability to critically review, interpret and apply the results from clinical studies to patient care, clinical pharmacy specialists have the potential to have a significant impact on stroke care delivery. There are numerous opportunities for clinical pharmacy specialists to become more extensively involved in the delivery of care to these high-risk patients. However, to-date there are few studies demonstrating the impact of clinical pharmacy specialists on outcomes of patients with stroke Stroke is the third leading cause of death in the United States (U.S.) and the most common life-threatening neurologic disorder.1 Stroke is a leading cause of long-term disability and results in significant individual and societal financial burdens. In 2006, stroke accounted for 1 of every 18 deaths and ischemic stroke accounted for 87% of all strokes.1 In the U.S., out of the approximately 795,000 people who develop a stroke each year, approximately 185,000 (23%) are recurrent events.1 After the first year, the average annual risk for recurrent stroke is 4%.2 Patients who survive at least 30 days after a first-ever stroke, have an average annual risk of death of 9.1%, much of the risk due to nonstroke cardiovascular disease.

Despite the evidence supporting the use of various therapeutic interventions within the ischemic stroke population, a significant proportion of patients continue to have uncontrolled risk factors and remain undertreated.26-30 A recent prospective study of more than 4933 high-risk patients reported that, as compared to patients with coronary artery disease, patients with cerebrovascular disease are undertreated and thus less likely to achieve blood pressure (45.3% vs. 57.3%; p<0.001) and lipid (19.4% vs. 30.5%; p<0.001) targets.28 Although the reasons for the so-called "treatment gap" have not been explored specifically within this population, data from studies within the coronary artery disease population suggest that provider, patient and health care system factors likely all contribute.

This will be the first, prospective, randomized study to evaluate the impact of a clinical pharmacist disease management program on both surrogate and clinical outcomes for patients with non-cardioembolic ischemic stroke.

This will be a randomized, controlled study comparing a clinical pharmacist-led disease management intervention by the Clinical Pharmacy Cardiac Risk Service (CPCRS) to usual care (UC).

DETAILED DESCRIPTION:
Aim 1: Conduct a randomized, controlled, study of a clinical pharmacist-led disease management intervention for patients with a history of non-cardioembolic ischemic stroke compared to usual care.

Hypothesis 1a: More patients in the clinical pharmacy specialist-led disease management group will achieve their lipid and blood pressure goals compared to the "Usual Care" group.

Hypothesis 1b: Fewer patients randomized to the clinical pharmacy specialist-led disease management group will have recurrent cardiovascular events or death compared to patients in the "usual care" group.

Hypothesis 1c: More patients with ischemic stroke will receive appropriate secondary prevention care using evidence-based medications in the intervention group compared to usual care.

All patients with ICD-9 codes 430.XX to 438.XX will be administratively identified from starting January 1, 2000 and administratively pulled into a HealthTrac®-Stroke registry. Each patient included in the registry will undergo a validation process to ensure stroke type and event dates are accurate. Staff at CPCRS will manually review the electronic medical record for each patient in the registry to ensure the ICD-9 code for stroke is accurate according to detailed procedures (Appendix I). Patients with history that indicates transient ischemic attack, subarachnoid hemorrhage, intracerebral hemorrhage, or cardioembolic stroke will be coded as "TIA" or "Hemorrhage" or "Cardioembolic" stroke, respectively, in the registry and not eligible for study screening or entry. Patients will be considered to have ischemic stroke if there is documentation in the medical record, hospital discharge summary or otherwise, indicating the patient had symptoms consistent with a stroke, for example but not limited to sudden numbness or weakness of the face, arm or leg, especially on one side of the body, sudden confusion, trouble speaking or understanding, sudden trouble seeing in one or both eyes, sudden trouble walking, dizziness, loss of balance or coordination, sudden, severe headache with no known cause) and/or imaging (MRI or CT scan) of clinically relevant brain lesions or there is documentation from a physician noting the patient has had a stroke.12 It is estimated that approximately 5200 patients will have validated stroke, of which 4200 will have ischemic stroke (both cardioembolic and non-cardioembolic) and approximately 2500 will have non-cardioembolic ischemic stroke. All eligible patients with a validated non-cardioembolic ischemic stroke diagnosis in the HealthTrac®-Stroke registry will be screened for study eligibility by study personnel.

Intervention (CPCRS) Group: The intervention will utilize clinical pharmacy specialists in CPCRS. The intervention will be similar to what is applied to patients with CAD. CPCRS will ensure patients have regular laboratory monitoring (i.e. lipids) and blood pressure measures, initiated on appropriate lipid-lowering and antihypertensive medications, and receive follow-up in a timely manner. CPCRS staff will order evidence-based lipid-lowering and/or antihypertensive medications, adjust doses, and order follow-up laboratory parameters, as necessary under pre-approved regional treatment protocols Patients will be monitored for medication adherence and adverse effects. Patients receive dietary, exercise, and smoking cessation counseling verbally and through mailing of pre-printed Kaiser Permanente approved, patient education pamphlets, as necessary per the discretion of the clinical pharmacy specialist. Patients requiring more intensive dietary counseling will be referred to appropriate resources offered at KPCO. Primary care providers will be informed of all medication initiations or dosage adjustments. The primary mode of communication between CPCRS and patients will be via telephone or e-mail through kp.org.

Usual Care: Patients randomized to Usual Care will continue to receive interventions/procedures they normally receive according to standard/usual care practices. Follow-up for Laboratories and Blood Pressure Values: Letters will be mailed to subjects in the Intervention group reminding him/her to have appropriate laboratories completed, as necessary, using standard CPCRS letters. Patients who fail to have laboratories drawn after 2 mailed reminder letters separated by 1-month will be marked "noncompliant" in the database and receive reminders every 6 months thereafter. For patients in the Usual Care group, no reminder letters will be sent. However for assessment of lipid and blood pressure control at 3 years (primary outcome) for both groups, reminder letters will be mailed, if necessary. All patients will be followed for 3 years from randomization or until the first occurrence of KPCO termination date, cardiovascular event, or death.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

All active KPCO non-institutionalized patients from the Denver/Boulder metropolitan area with a validated non-cardioembolic ischemic stroke diagnosis within the past 5 years who:

Are ≥18 years of age at the time of informed consent, and Are Eligible for CPCRS enrollment, and Have uncontrolled blood pressure (the most recent value >130/80 mmHg noted in the medical record), and/or Have last LDL-C, within the previous 365 days, that is ≥100 mg/dL.

Exclusion Criteria:

Patients will be excluded if:

* 85 years of age at the time of consent, Have transient ischemic attacks, subarachnoid hemorrhage,intracerebral hemorrhage, or cardioembolic stroke as their only validated stroke history, Die within 30 days of stroke, Are already followed by the Clinical Pharmacy Cardiac Risk Service (CPCRS). These patients either have a history of coronary artery disease (acute MI, CABG, percutaneous coronary interventions, and/or coronary catheterizations), are at high-risk for CAD as determined by the cardiologist, or have peripheral arterial disease, Have a diagnosis of dementia or a terminal illness in which the life expectancy is <3 years per the discretion of the primary care provider, Have notation in the medical record of memory issues or other conditions which, based on the judgment of study staff, suggest that the patient may not be able to provide informed consent, Are pregnant or breast-feeding, or Do not consent to participate Currently listed on the "Do Not Call List"

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2010-07; Primary Completion 2016-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the proportion of patients in each group who attain recommended LDL-C and BP goals 3 years after randomization. | 5 years
  The outcome measures selected for the study are based on AHA/ASA guidelines for prevention of stroke in patients with ischemic stroke or transient ischemic attack.19,20 The surrogate measures to be evaluated are the "ABCs" which include Antiplatelet/antithrombotic therapy, Blood pressure control, Cholesterol control, and Smoking cessation. These variables will be evaluated at various time points during the study in part to evaluate the CPCRS processes of care for attaining surrogate measures in the short-term and maintenance of these outcomes long-term compared to Usual Care. Surrogate outcome measures will be evaluated at 1 and 3 years after randomization.
  The LDL-C goal will be <100 mg/dL for all patients as recommended by clinical practice guidelines.19,20 The proportion of patients with an LDL-C <70 mg/dL in each group will also be reported

SECONDARY OUTCOMES:
Major cardiovascular events | 5 years
  Cardiovascular events will include fatal or non-fatal stroke, coronary events, or revascularization procedures. Stroke will include either ischemic or hemorrhagic. Coronary events will include acute myocardial infarction ± percutaneous coronary intervention, percutaneous coronary intervention, or coronary artery bypass graft surgery (CABG) surgery. Revascularization procedures include percutaneous coronary intervention, coronary artery bypass graft surgery (CABG) surgery, carotid endarterectomy, interarterial stent insertion. Events will be captured administratively using ICD-9 and/or CPT codes and will be reviewed by individuals blinded the randomization scheme.
Hospitalizations | over study period
  Hospitalizations for any reason will be collected over the study period for all patients.
Death | over study period
  : Death will be captured through KPCO administrative databases. Cause of death will be determined by death certificates and classified as any-cause or cardiovascular. If not cause of death is noted on the death certificate, the cause will be assumed to be cardiovascular. Cardiovascular deaths will include death from cardiac causes, ruptured aortic aneurysm, or peripheral vascular disease. Sudden deaths will be regarded as cardiovascular unless an alternative explanation is documented.

OTHER OUTCOMES:
Tertiary Outcomes | over study period
  Tertiary outcome measures will describe the effectiveness and safety of the intervention as compared to Usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Kari L Olson, PharmD, Principal Investigator — Kaiser Permanente
Locations (1):
- Clinical Pharmacy Specialist, Clinical Pharmacy Cardiac Risk Service - Kaiser Permanente of Colorado, Aurora, Colorado, United States